CLINICAL TRIAL: NCT06528093
Title: A First-in-human Open Label Phase Ia/Ib, Multicenter/Multiregional, Dose Escalation Study of BI 765883 Administered Intravenously as Monotherapy and in Combination With Gemcitabine and Nab-paclitaxel in Unselected Patients With Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC) or Patients With PDAC Who Have Relapsed After Post-surgery Adjuvant Therapy
Brief Title: A Study to Find a Suitable Dose of BI 765883 and to Test Whether it Helps People With Advanced Pancreatic Cancer When Taken Alone or Together With Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Primary endpoint not met
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1505-0001; 2023-508998-85-00 (Registry Identifier: CTIS); U1111-1300-7624 (Other: WHO)
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BI 765883 escalation arm (Experimental): phase Ia
  Interventions: Drug: BI 765883
- BI 765883 + gemcitabine + nab-paclitaxel escalation arm (Experimental): phase Ia
  Interventions: Drug: BI 765883; Drug: gemcitabine; Drug: nab-paclitaxel
- BI 765883 + gemcitabine + nab-paclitaxel expansion arm (Experimental): phase Ib
  Interventions: Drug: BI 765883; Drug: gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: BI 765883 — BI 765883
Drug: gemcitabine — gemcitabine
  Arms: BI 765883 + gemcitabine + nab-paclitaxel escalation arm; BI 765883 + gemcitabine + nab-paclitaxel expansion arm
Drug: nab-paclitaxel — nab-paclitaxel
  Arms: BI 765883 + gemcitabine + nab-paclitaxel escalation arm; BI 765883 + gemcitabine + nab-paclitaxel expansion arm

SUMMARY:
This study is open to adults with advanced pancreatic cancer for whom previous treatment was not successful or no treatment exists.

The purpose of this study is to find the highest dose of BI 765883 that people with advanced pancreatic cancer can tolerate when taken alone or together with chemotherapy. Another purpose is to check whether BI 765883 helps people with advanced pancreatic cancer. In this study, BI 765883 is given to humans for the first time.

Participants receive either BI 765883 alone or BI 765883 in combination with chemotherapy. Participants can stay in the study as long as they benefit from treatment and can tolerate it. At study visits, doctors collect information on any health problems of the participants and check the severity of participants' cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
2. Of legal adult age (according to local legislation) at screening
3. Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be willing and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.
4. Histologically or cytologically confirmed Pancreatic ductal adenocarcinoma (PDAC)
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
6. Life expectancy ≥3 months in the opinion of the investigator
7. Archived tumor tissue from a tissue core biopsy (e.g. paraffin-embedded formalin-fixed tissue blocks), OR fresh tumor tissue available for retrospective biomarker analysis; in both cases, a minimum of at least two core needle biopsies (18 gauge or greater) is required. Only non-significant risk procedures per the investigator's judgment will be used to obtain any biopsies specified in this study in cases where a fresh tumor biopsy is required.
8. Patients with at least 1 target lesion that can be accurately measured per RECIST version 1.1 Further inclusion criteria apply.

Exclusion Criteria:

1. Previous exposure to trial drug (BI 765883)
2. Any prior gemcitabine and/or paclitaxel therapy (for combination therapy cohorts)
3. Known hypersensitivity to the study medications or their excipients (including gemcitabine and nab-paclitaxel)
4. Any contraindications to gemcitabine or nab-paclitaxel according to the current approved local labels (combination therapy)
5. Currently enrolled in another investigational device or drug trial, or less than 28 days since ending another investigational device or drug trial(s) or receiving other investigational treatment(s)
6. Any serious concomitant disease or medical condition affecting compliance with trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug, such as neurologic, psychiatric, infectious disease, active ulcers (gastrointestinal tract, skin), inflammatory bowel disease or bowel infection, or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the Investigator, would make the patient inappropriate for entry into the trial.
7. Prior radiotherapy or systemic therapy within 14 days prior to treatment start
8. History or presence of cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of ≥III or IV, unstable angina or poorly controlled arrhythmia which are considered as clinically relevant by the Investigator Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities (DLTs) in the maximum tolerated dose (MTD) evaluation period | Up to 28 days (2 treatment cycles)
  phase Ia
Confirmed objective response (OR) | Up to 350 days (25 treatment cycles)
  phase Ib

SECONDARY OUTCOMES:
Objective response (OR) | Up to 350 days (25 treatment cycles)
  phase Ia
Recommended dose for expansion (RDE) for BI 765883 in combination with gemcitabine and nab-paclitaxel | Up to 28 days (2 treatment cycles)
  phase Ia
Frequency and severity of AEs according to the Common Terminology Criteria for Adverse Events (CTCAE) | Up to 350 days (25 treatment cycles)
  phase Ia and phase Ib
Maximum measured concentration of the analyte in serum (Cmax) | Up to 350 days (25 treatment cycles)
  phase Ia and phase Ib
Area under the serum concentration time curve of the analyte (AUC0-t) | Up to 350 days (25 treatment cycles)
  phase Ia and phase Ib
Progression-free survival (PFS) | Up to 350 days (25 treatment cycles)
  phase Ib
Duration of response (DOR) | Up to 350 days (25 treatment cycles)
  phase Ib

CONTACTS AND LOCATIONS:
Locations (17):
- United States (5):
  - HealthONE, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists-Sarasota-61670, Sarasota, Florida
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- France (3):
  - CTR Leon Berard, Lyon
  - CTR Eugène Marquis, Rennes
  - INS Gustave Roussy, Villejuif
- Germany (3):
  - Universitätsklinikum Hamburg, Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum der Universität München AÖR, München
- Japan (2):
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - National Cancer Center Hospital, Tokyo, Chuo-ku
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com